CLINICAL TRIAL: NCT04716439
Title: Effect of Total Intravenous Anesthesia (TIVA) With Magnesium Sulfate on Intra-Operative Neuromonitoring (IONM) in Patients Undergoing Spine Surgery
Brief Title: Effect of TIVA With Magnesium Sulfate on IONM in Patients Undergoing Spine Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: King Khalid University Hospital (Other)
Responsible Party: Principal Investigator, Essam M. Manaa (MD), Assistant Professor & Consultant, King Khalid University Hospital
Other Study IDs: E-20-4965
Record Dates: First submitted 2021-01-11; First posted 2021-01-20 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Spine Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- magnesium sulfate effect on IONM reading in spine surgery: one group receives magnesium other do not
  Interventions: Procedure: Spine Surgery

INTERVENTIONS:
Procedure: Spine Surgery — spine decompression and fixation

SUMMARY:
Anesthesia for neurosurgery requires balancing deep and effective anesthesia as well as postoperative analgesia versus the risks of delayed recovery and postoperative respiratory depression. This randomized placebo-controlled, double-blind study was designed to evaluate the effect of magnesium sulfate on the total anesthetic and analgesic consumption using the clinical parameters in addition to the effect on IONM reading.

DETAILED DESCRIPTION:
Objectives:

1. Decrease anesthetic consumption
2. Decrease use of muscle relaxants
3. Decrease analgesic consumption
4. Excellent recovery

Patients & Methods:

* 2 groups (total 50) Randomized Controlled Double Blind (RCDB) Study
* Propofol + remifentanil + saline (Control = C group)
* Propofol + remifentanil + Mgso4 (Magnesium = M group)
* Adult Spine decompression and fixation After getting the Institutional Review Board (IRB) approval, This randomized controlled double blind study includes 2 groups of patients (each group 25) will be enrolled in the study. All patients undergo spine decompression and fixation surgery

Induction:

All patients in the study will receive iv fentanyl 2 mic/kg + propofol 2mg/kg and endotracheal intubation will be facilitated with rocuronium 0.60 mg/ kg. Then anesthesia will be maintained using total intravenous anesthesia with propofol (6-9 mg/kg/hr) + remifentanil (0.03-0.05 mic / kg/ min) Group 1 (C group) : Receive 10 mg/kg /hr 0.9% Normal Saline Group 2 (M group) : Receive 10 mg/kg/hr Magnesium Sulfate

Monitoring:

1. IONM
2. train-of-four (TOF)
3. bispectral index (BIS)

Measurements:

1. IO Anesthetic Consumption
2. IO Hemodynamics
3. somatosensory evoked potential (SSEP), motor evoked potential (MEP), TOF, BIS Readings
4. PO visual analogue scale (VAS) (24hours)
5. PO Morphine Consumption (24hours)

ELIGIBILITY:
Inclusion Criteria:

* Adult Patients Undergoing Spine Surgery

Exclusion Criteria:

1. Renal Impairment
2. Liver Cell failure
3. Heart Block

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult ASA 1OR 2
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
IONM Reading | 1- baseline 2-during surgery 3-immediately after surgery
  Reading the effect on the intraoperative neuromonitoring either motor or sensory evoked potential

SECONDARY OUTCOMES:
Blood Pressure | 1- baseline 2-during surgery 3-immediately after surgery 4- every one hour postoperative till 24 hours
  Systolic, Diastolic and Mean (mmHg)
Heart Rate | 1- baseline 2-during surgery 3-immediately after surgery 4- every one hour postoperative till 24 hours
  beats/min
Morphine Consumption | Over 24 hours postoperative
  Total morphine consumed over 24 hours in mg
Pain Score | Over 24 hours postoperative
  11 Visual Analogue Scale (VAS) with 10 is the worst and 0 is the least

CONTACTS AND LOCATIONS:
Overall Officials: ESSAM M MANAA, MD, Principal Investigator — Assistant Professor and Consultant, Anesthesia Department, Faculty of Medicine, KKUH, KSU, Riyadh, Saudi Arabia
Locations (1):
- Anesthesia Department, Faculty of Medicine, King Khalid University Hospital, King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No